CLINICAL TRIAL: NCT06962410
Title: Application of a Hybrid Closed-Loop Artificial Pancreas System in Patients With Diabetes After Kidney Transplantation: An Open-Label, Randomized Controlled Trial
Brief Title: Hybrid Closed-Loop in Diabetes Post-Kidney Transplant: A Randomized Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-2025-027
Record Dates: First submitted 2025-04-22; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus Patients With Kidney Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Insulin Pump and CGM Group (Experimental): Calculate the total daily insulin requirement based on the patient's weight at a rate of 0.2-0.4 U/（kg·d）, and allocate it to premeal doses according to the patient's specific condition. Monitor blood glucose levels using a continuous glucose monitoring system, combined with five daily capillary blood glucose tests (fasting, 2 hours after breakfast, 2 hours after lunch, 2 hours after dinner, and before bedtime). Adjust the insulin dosage according to the patient's blood glucose levels until the target range is achieved.
  Interventions: Other: Hybrid Closed-Loop Artificial Pancreas System
- Hybrid Closed-Loop Artificial Pancreas with CGM Group (Placebo Comparator): The hybrid closed-loop artificial pancreas group: An open-source hybrid closed-loop system was used with ultra-short-acting insulin (Novo Nordisk A/S, Denmark; Approval No.: J20050097; Spec.: 3 mL: 300 U). The total daily insulin dose was calculated at 0.2-0.4 U/(kg·d) based on patient weight. The system automatically adjusted the basal rate based on blood glucose levels. Physicians prescribed bolus doses based on prior experience and glucose readings, which nurses manually entered into the AAPS software. Continuous glucose monitoring (CGM) was used, with five daily fingerstick capillary blood glucose tests for correction (fasting, 2 hours post-breakfast, lunch, dinner, and before sleep). The AAPS system had a low glucose prediction suspend feature, pausing basal infusion when glucose was predicted to drop below 4.4 mmol/L until it returned to a safe range. An alarm threshold was set at <3.9 mmol/L with a loud volume to awaken patients during deep sleep.
  Interventions: Other: Hybrid Closed-Loop Artificial Pancreas System

INTERVENTIONS:
Other: Hybrid Closed-Loop Artificial Pancreas System — The pump was loaded with ultra-short-acting insulin (Manufacturer: Novo Nordisk A/S, Denmark; Approval Number: National Drug Approval No. J20050097; Specification: 3 mL: 300 U). The total daily insulin requirement was calculated at 0.2-0.4 U/(kg·d) based on the patient's weight. During operation, the system automatically adjusted the basal rate according to the blood glucose level. After the physician issued a large-dose order based on previous treatment experience and blood glucose conditions, the nurse manually entered the large-dose treatment instruction in the AAPS software.

SUMMARY:
Objective: To evaluate the short-term blood glucose control effect of the closed-loop system combined with a regular insulin pump and continuous glucose monitoring (CGM) in hospitalized patients with diabetes after kidney transplantation, explore its clinical application value, and provide precise and personalized blood glucose management plans. Methods: A clinical comparative study will be conducted. This will be the first study focusing on hospitalized patients with diabetes after kidney transplantation. The advanced closed-loop system technology will be introduced. Expected Results: The study aims to fill the gap in this field, offer new ideas and solutions for clinical blood glucose management of these patients, and promote the development of diabetes treatment technologies by comparing the short-term blood glucose control effects of the closed-loop system and the regular insulin pump combined with CGM.

DETAILED DESCRIPTION:
Based on the difficulty in blood glucose control for patients with diabetes after kidney transplantation and the insufficiency of previous studies, this research intends to conduct a clinical comparative study to evaluate the short-term blood glucose control effect of the closed-loop system combined with a regular insulin pump and CGM in hospitalized patients with diabetes after kidney transplantation, explore its clinical application value in this patient group, and provide more precise and personalized blood glucose management plans for them. This study will be the first to focus on patients with diabetes after kidney transplantation, especially the hospitalized ones, filling the gap in this field. Meanwhile, by introducing the most advanced closed-loop system technology, it aims to offer new ideas and solutions for the clinical blood glucose management of these patients. Through the comparative analysis of the short-term blood glucose control effects of the closed-loop system and the regular insulin pump combined with CGM, this research aims to provide more precise and personalized treatment strategies for patients with diabetes after kidney transplantation and promote the further development of diabetes treatment technologies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 70 years;
* Meets the diagnostic criteria in the "Guidelines for Prevention and Control of Diabetes in China (2024 Edition)": A patient can be diagnosed with diabetes if he/she presents typical symptoms of diabetes (including polydipsia, polyuria, polyphagia, and unexplained weight loss) and meets one of the four criteria: ① random blood glucose ≥ 11.1 mmol/L; ② fasting blood glucose ≥ 7.0 mmol/L; ③ 2 - hour post - load blood glucose during an oral glucose tolerance test ≥ 11.1 mmol/L. For patients without typical symptoms, the diagnosis requires two abnormal test results obtained either simultaneously or at two different time points.
* Able to correctly use insulin pumps and CGM devices, and has certain learning and operational abilities;
* Agrees to participate in the study and signs the informed consent form.

Exclusion Criteria:

* The patient has experienced acute diabetic complications within the past month, such as diabetic ketoacidosis, hyperglycemic hyperosmolar coma, etc.
* The patient has severe symptoms of hypoglycemic intolerance.
* The patient has skin diseases such as rashes and prurigo, or abnormal coagulation function.
* The patient has diseases related to glucose metabolism, such as uncontrolled hyperthyroidism, uncontrolled hypothyroidism, Cushing's syndrome, etc.
* The patient has severe diseases of the liver, kidneys, gastrointestinal tract, hematopoietic system, brain, circulatory system, etc.
* Patients with malignant tumors (including solid tumors and hematological malignancies).
* The patient has impaired consciousness or mental illness, lacks self-control, and is unable to express clearly.
* Lactating women, pregnant women, or women who plan to become pregnant during the trial period.
* The patient is allergic to the drugs involved in the clinical diagnosis and treatment plan.
* The patient is currently using other closed-loop systems.
* Populations not suitable for conventional insulin pump therapy and contraindications.
* The patient has known or suspected insulin allergy, or is allergic to adhesive tape, insulin pumps, or CGM devices.
* Other situations where the investigator deems the patient unfit to participate in the clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Days Required to Achieve 70% TIR | 2 years
  The number of days required for a patient to achieve a Time in Range (TIR) of 70%, where TIR is defined as the percentage of time that blood glucose levels are maintained within the target range of 3.9-10.0 mmol/L. This metric is calculated using the formula: TIR = (Time in Range / Total Time) × 100%.
The blood glucose target achievement rate during 5×24 hours of treatment. | 2 years
  The blood glucose target achievement rate during 5×24 hours of treatment refers to the percentage of time that a patient's blood glucose levels are maintained within the target range (typically 3.9-10.0 mmol/L) over a continuous 5-day (120-hour) treatment period. This metric is used to assess the effectiveness of the treatment regimen in maintaining stable blood glucose levels over an extended period.

SECONDARY OUTCOMES:
Blood Glucose Target Achievement Rate (TAR) | 2 years
  In the absence of hypoglycaemia, the fasting blood glucose is less than 7.0 mmol/L, and the 2 - h postprandial blood glucose is less than 10.0 mmol/L. The blood glucose target achievement rate within one week of intensive insulin therapy is calculated as: Blood Glucose Target Achievement Rate = (Number of Patients with Blood Glucose under Control / Total Number of Patients) × 100%.
Time Below Range (TBR) ，Time Above Range (TAR) | 2 years
  Time Below Range (TBR) is the percentage of time that blood glucose is below the target range (<3.9 mmol/L). It's calculated as TBR = (Time with blood glucose <3.9 mmol/L / Total time) × 100%. Time Above Range (TAR) is the percentage of time that blood glucose is above the target range (>10.0 mmol/L). It's calculated as TAR = (Time with blood glucose >10.0 mmol/L / Total time) × 100%.
Hypoglycemia incidence | 2 years
  Hypoglycemia incidence rate refers to the frequency of blood glucose levels falling below a predefined threshold, typically <3.9 mmol/L, during a specified monitoring period. It reflects how often hypoglycemic events occur in relation to the total monitoring time or number of patients monitored.
Blood Glucose Variability (IQR) | 2 years
  The 25th and 75th percentile values of blood glucose fluctuations (Interquartile Range, IQR).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No
If there is a need to use data, please contact the person in charge and follow the relevant procedures to achieve data sharing. Without permission, do not use the data directly.